CLINICAL TRIAL: NCT01977833
Title: Effects of Meal Timing on Postprandial Glucose, Insulin and GLP-1 Responses After Breakfast Lunch and Dinner in Patients With Type 2 Diabetes
Brief Title: Meal Timing on Postprandial Glucose, Insulin and GLP-1 in Type 2 Diabetes
Acronym: GLP-1inT2D
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel Aviv University (Other)
Collaborators: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Daniela Jakubowicz, Professor Daniela Jakubowicz MD, Tel Aviv University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0145-13-WOMC
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-10

CONDITIONS: Type 2 Diabetes
Keywords: BTdiet; Dtdiet; High Calorie Breakfast diet (BTdiet); High Calorie Dinner diet (DTdiet)
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Calorie Breakfast (BTdiet) (Experimental): High Calorie Breakfast (BTdiet): The subject will consume High caloric breakfast, average lunch and reduced in calories dinner (BTdiet)
  Interventions: Other: High Calorie Breakfast (BTdiet)
- High Calorie Dinner (DTdiet) (Active Comparator): High Calorie Dinner (DTdiet): The subject will consume High caloric dinner, average lunch and reduced in calories breakfast (DTdiet)
  Interventions: Other: High Caloric Dinner (DTdiet)

INTERVENTIONS:
Other: High Calorie Breakfast (BTdiet) — High Caloric Breakfast Test Diet (BTdiet): in which the majority of energy load will be consumed in the morning and with reduced dinner
  Arms: High Calorie Breakfast (BTdiet)
Other: High Caloric Dinner (DTdiet) — High Caloric Dinner (DTdiet): resembling a skipping breakfast plan, in which the majority of energy load will be consumed in the evening with minimal caloric content at breakfast
  Arms: High Calorie Dinner (DTdiet)

SUMMARY:
Enhanced insulin and GLP-1 postprandial response after morning meal versus evening meal, might be underlying explanation of the beneficial effect of eating breakfast with reduced dinner vs skipping breakfast on glycemic control and HbA1c in T2D patients.

To test this hypothesis and clarify whether glucose, insulin and GLP-1 postprandial responses are different in the morning vs. in the afternoon, the investigators will compare in T2D subjects in random order and in two separate days: the glucose, insulin and GLP-1 postprandial responses after breakfast, lunch and dinner with 2 isocaloric meal plans or test diets, that differ in meal timing distribution The investigators hypothesize that GLP-1 and insulin response after high calorie breakfast will be higher in comparison to GLP-1 and insulin response after identical meal at evening

DETAILED DESCRIPTION:
The endogenous circadian (24-h) timing system, synchronized by light/dark cycle in the master circadian clock in the suprachiasmatic nuclei and by meal timing in the peripheral clock genes; plays a significant role in regulating sleep/wake and feeding behavior, body weight as well as glucose and lipid metabolism.

Circadian misalignment, involving sleep/wake and meal timing schedules 12 h out of phase from their habitual times resulted in elevated blood pressure and increased postprandial glucose and insulin levels. Animal models of circadian misalignment specially breakfast skipping are associated with alteration in the expression pattern of clock genes such as Clock, Bmal1, Cry1, and Per2 in the liver and fat cells. These changes resulted in a predisposition to obesity and type 2 diabetes (T2D). This may also explain why evening or night eating is often associated with weight gain and obesity.

Breakfast skipping has been consistently associated with increased, visceral adiposity, higher BMI and waist circumference, insulin resistance, dyslipidemia and with T2D despite having less total daily caloric intake.

A recent population-based studies have found that participants with an evening preferences (late chronotype) that involves breakfast skipping, have 2.5 times risk of developing T2D, even after adjustment for body mass index (BMI) (12).

Breakfast skipping and greater percentage of their daily caloric intake at dinner was associated with higher fasting plasma glucose levels, and poorer glycemic control compared with earlier chronotypes even after adjusting for BMI (11,20,21). Recently was documented that in T2D patients, breakfast skipping was associated was associated with a 10.8% increase in HbA1C of its original value, even after adjusting for age, sex, race, BMI, number of diabetes complications, insulin use, depressive symptoms, perceived sleep debt, and percentage of daily caloric intake at dinner. This significant difference in HbA1C levels between breakfast skippers and breakfast eaters in patients with T2D, highlights the potential impact of the meal timing on the course of the disease.

More recently the investigators documented that compared to a conventional diet, a high caloric intake in the breakfast and reduced dinner resulted in significant reduction of HbA1c in T2D individuals.

The existence of diurnal variation in glucose tolerance in healthy and in subjects with T2D has been suspected for decades, with reports showing that glucose tolerance decreases progressively throughout the day with insulin sensitivity reaching a nadir in the evening. The reduction of glucose tolerance in the evening, seems to be a results from a combination of reduced glucose utilization, decreased insulin sensitivity, and inappropriately low insulin secretion and action, which highlights the importance of meal timing in glucose metabolism.

It is known that insulin response to meal ingestion is more rapid in the morning than in the afternoon and specifically the early (30 or 45 min) insulin secretion after oral glucose or meal ingestion is significantly higher in the morning than in the evening. A possible explanation for the more rapid glucose clearance from the circulation in the morning is because the early insulin response is important for rapid reduction in hepatic glucose output after meal ingestion.

Recently was shown that the enhanced early (30-min) insulin secretion after morning meal vs. afternoon, was accompanied by a correspondingly faster incretin total GLP-1 and intact GLP-1 hormone response in the morning specially during the first 30 min after ingestion. The association was consistent and also supports the prediction that higher GLP-1 levels after morning meal would result in a higher potentiation of β-cell function.

This diurnal pattern of enhanced insulin and GLP-1 response after morning meal versus in the evening, might be underlying explanation of the beneficial effect of eating breakfast with reduced dinner vs skipping breakfast on glycemic control and HbA1c in T2D patients.

To test this hypothesis the investigators will compare in random order and in two separate days: the glucose, insulin and GLP-1 postprandial responses after breakfast, lunch and dinner with 2 isocaloric meal plans or test diets, that differ only in meal timing distribution

1. High caloric breakfast, average lunch and reduced dinner (BTdiet) and
2. High caloric dinner, similar lunch and reduced breakfast (DTdiet)

ELIGIBILITY:
Inclusion Criteria:

1. Type 2 diabetes patients
2. HbA1C > 7%
3. Duration of diabetes: 0.5 to 10 years
4. Subjects ≥ 30 and ≤70 years of age
5. BMI: 22 to 35 kg/m2
6. Diet controlled diabetic. Only treatment with metformin will be allowed
7. Normal liver and kidney function
8. Normal thyroid function
9. Acceptable health beside diabetes based on interview, medical history, physical examination, and laboratory tests
10. Stable physical activity pattern during the three months immediately preceding study
11. Usually wakes up between 06:00 and 07:00 and goes to sleep between 22:00 and 24:00.
12. No shift work within 5 years of the study
13. Did not cross time zones within 1 month of the study
14. Read and understood the informed consent form and signed it voluntarily

Exclusion Criteria:

1. Type 1 diabetes
2. Clinically significant pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious, malignant disease
3. Abnormal liver function tests defined as an increase by a factor of at least 2 above the upper normal limit of alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST)
4. Pregnancy or lactation
5. Illicit drug abuse or alcoholism
6. Treatment with antidiabetic drugs, insulin or GLP-1 analogs
7. Subjects taking anoretic drugs during the month immediately prior to study
8. Subjects on steroid treatment
9. Those with eating disorders
10. Subjects after bariatric surgery, will be excluded

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-10; Primary Completion 2013-12 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Postprandial GLP-1 plasma levels, after breakfast,lunch and dinner meal test | During 3 hours after breakfast, lunch and dinner meal challange
  All Type 2 diabetic participants will be randomly assigned to one of 2 isocaloric diet sequences that will differ in the meal timing distribution. The diets will be tested in two separate occasions during a curse of a single day (test day) in which postprandial plasma GLP-1 levels during 3 hours after breakfast, lunch and dinner meal challenge will be measured

SECONDARY OUTCOMES:
Postprandial Plasma Glucose levels after breakfast, lunch and dinner meal challenge | Postprandial Plasma Glucose levels during 3 hours after breakfast, lunch and dinner meal challenge
  All Type 2 diabetic participants will be randomly assigned to one of 2 isocaloric diet sequences that will differ in the meal timing distribution. The diets will be tested in two separate occasions during a curse of a single day (test day) in which postprandial plasma Glucose levels during 3 hours after breakfast, lunch and dinner meal challenge will be measured

OTHER OUTCOMES:
Postprandial Insulin plasma levels, after breakfast,lunch and dinner meal test | During 3 hours, after breakfast,lunch and dinner meal test
  All Type 2 diabetic participants will be randomly assigned to one of 2 isocaloric diet sequences that will differ in the meal timing distribution. The diets will be tested in two separate occasions during a curse of a single day (test day) in which postprandial plasma Insulin levels during 3 hours after breakfast, lunch and dinner meal challenge will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Jakubowicz, Principal Investigator — E. Wolfson Medical Center. Tel Aviv University
Locations (1):
- Diabetes Unit E. Wolfson Medical center, Holon, Tel Aviv, Israel

REFERENCES:
- [Derived] Jakubowicz D, Wainstein J, Ahren B, Bar-Dayan Y, Landau Z, Rabinovitz HR, Froy O. High-energy breakfast with low-energy dinner decreases overall daily hyperglycaemia in type 2 diabetic patients: a randomised clinical trial. Diabetologia. 2015 May;58(5):912-9. doi: 10.1007/s00125-015-3524-9. Epub 2015 Mar 1. PMID 25724569